CLINICAL TRIAL: NCT05292612
Title: Chinese Internet-delivered Cognitive Therapy for Social Anxiety Disorder in Hong Kong: A Randomised Controlled Noninferiority Trial to Compare Clinician Versus Coach Guidance
Brief Title: CvC-SAD (Clinician vs Coach)Self-help Versions in a RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Patrick Wing-Leung LEUNG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022.086-T
Record Dates: First submitted 2022-02-23; First posted 2022-03-23 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard therapist-guided iCT-SAD vs. Waitlist (Experimental): to examine if standard iCT-SAD delivered in Chinese is superior to waitlist.
  participants in the experimental group would receive iCBT(C&W) for SAD under the guidance of trained therapist.
  Interventions: Behavioral: iCBT(C&W) for SAD
- Guided self-help iCT-SAD vs. Waitlist (Experimental): to examine if guided self-help iCT-SAD delivered in Chinese is superior to waitlist.
  participants in the experimental group would receive iCBT(C&W) for SAD under the guidance of trained coaches.
  Interventions: Behavioral: iCBT(C&W) for SAD
- Standard therapist-guided iCT-SAD vs. Guided self-help iCT-SAD (Experimental): to examine if guided self-help iCT-SAD is noninferior to standard iCT-SAD.
  participants would be randomised into two groups. one group of participants would receive iCBT(C&W) for SAD under the guidance of trained therapist while the other group of participants would receive iCBT(C&W) for SAD under the guidance of trained coaches.
  Interventions: Behavioral: iCBT(C&W) for SAD

INTERVENTIONS:
Behavioral: iCBT(C&W) for SAD — iCBT(C&W) for SAD implements all the key procedures of the face-to-face treatment. Patients are guided through the treatment by using secure messaging and regular telephone or webcam calls. The treatment comprises a series of online modules, each of which includes educational texts, patient testimonies, video illustrations, case examples, questionand- answer boxes, monitoring sheets, behavioural experiments and other homework assignments.

SUMMARY:
Background:

Social Anxiety Disorder (SAD) is a common mental problem, where people experience severe and disabling anxiety about social situations and interactions. It is highly prevalent world-wide and in Hong Kong, causing significant suffering/distress. While evidence-based interventions exist, e.g., cognitive behavioural therapy (CBT), there will be not enough trained therapists to meet the treatment demand so that the majority of the SAD patients receive no treatment. Internet-based therapies may offer a solution, given that they deliver treatment more cost-efficiently by requiring lesser therapist time so that more patients can be treated with the same therapist resources. One UK internet-based CBT protocol for SAD, iCBT(C&W), shows high efficacy and efficiency in initial UK and Hong Kong trials with Englishspeaking patients.

Objectives:

1. To develop and confirm the efficacy of a Chinese-language version of iCBT(C&W), administered by clinical psychologists in standard therapist-guided format.
2. To develop an even more cost-efficient new self-help format with some minimal 'coaching' performed by trained psychology bachelor-level graduates - its efficacy expected as 'noninferior' to that of the therapist-guided format.

Overall design:

Three-arm parallel group randomised controlled noninferiority trial: Standard therapist-guided iCT-SAD vs. Guided self-help iCT-SAD vs. Waitlist

Method:

The iCBT(C&W) protocol will be translated into Chinese. Approximately 110 Chinese adults with SAD will be recruited in Hong Kong and randomised into one of two treatment conditions, therapist-guided versus self-help. The treatment lasts 14 weeks. The primary outcome measure will be Liebowitz Social Anxiety Scale (self-report version).

ELIGIBILITY:
Inclusion

* Meets DSM-5 criteria for SAD (SAD must be generalised, not the 'performance only' subtype)
* Considers SAD their main problem
* Age 18 or over (no upper age limit)
* No current psychotropic mediation, or on a stable dose for at least two months without improvement, and willing to remain at this dose throughout trial
* Participant agrees not to start any other forms of treatment during the trial
* Chinese resident of Hong Kong
* Proficient in written traditional Chinese and spoken Cantonese
* Internet access from home

Exclusion

* current or past psychosis, bipolar disorder, or borderline personality disorder
* active suicidality
* 'Moderate' or 'Severe' Alcohol Use Disorder or Substance Use Disorder (based on DSM-5)
* No current or previous CBT for SAD (defined as at least 5 sessions, and including an exposure component), including internet-CBT studies
* Not another current emotional problem that is the participant's main concern (Participant must not be largely absorbed in another emotional problem, for which it would be unethical not to address as a priority)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale, Self-report version (LSAS) | through study completion, an average of 14 weeks
  LSAS consists of twenty-four items to assess individual's fear and avoidance towards different social interactions and performance situations. A total of six subscale scores could be obtained in LSAS, including the total fear, fear of social interactions, fear of performance situations, total avoidance, avoidance of social interactions, and avoidance of performance situations.
Liebowitz Social Anxiety Scale, Self-report version (LSAS) | at 3-month post-treatment follow-up
  LSAS consists of twenty-four items to assess individual's fear and avoidance towards different social interactions and performance situations. A total of six subscale scores could be obtained in LSAS, including the total fear, fear of social interactions, fear of performance situations, total avoidance, avoidance of social interactions, and avoidance of performance situations.
Liebowitz Social Anxiety Scale, Self-report version (LSAS) | at 9-month post-treatment follow-up
  LSAS consists of twenty-four items to assess individual's fear and avoidance towards different social interactions and performance situations. A total of six subscale scores could be obtained in LSAS, including the total fear, fear of social interactions, fear of performance situations, total avoidance, avoidance of social interactions, and avoidance of performance situations.

SECONDARY OUTCOMES:
Patient Health Questionnaire-Depression Scale (PHQ-9) | through study completion, an average of 14 weeks
  PHQ-9 consists of nine items that captures the criterion symptoms of DSM-5 major depressive disorder
Patient Health Questionnaire-Depression Scale (PHQ-9) | at 3-month post-treatment follow-up
  PHQ-9 consists of nine items that captures the criterion symptoms of DSM-5 major depressive disorder
Generalized Anxiety Disorder-7 (GAD-7) | through study completion, an average of 14 weeks
  GAD-7 consists of seven items that captures the criterion symptoms of DSM-5 common anxiety disorders
Generalized Anxiety Disorder-7 (GAD-7) | at 3-month post-treatment follow-up
  GAD-7 consists of seven items that captures the criterion symptoms of DSM-5 common anxiety disorders
Work and Social Adjustment Scale (WSAS) | through study completion, an average of 14 weeks
  WSAS consists of five items that measure participants' perceived functional impairment incurred by their presenting psychiatric problem (which, in this study, refers to SAD)
Work and Social Adjustment Scale (WSAS) | at 3-month post-treatment follow-up
  WSAS consists of five items that measure participants' perceived functional impairment incurred by their presenting psychiatric problem (which, in this study, refers to SAD)
Social Phobia Weekly Summary Scale (SPWSS) | through study completion, an average of 14 weeks
  SPWSS is a five-item self-report questionnaire on social anxiety, social avoidance, self-focused versus external-focused attention, anticipatory processing, and post-event rumination.
Social Phobia Weekly Summary Scale (SPWSS) | at 3-month post-treatment follow-up
  SPWSS is a five-item self-report questionnaire on social anxiety, social avoidance, self-focused versus external-focused attention, anticipatory processing, and post-event rumination.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Leung, Prof., Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No